CLINICAL TRIAL: NCT00584506
Title: Computer Aided Evaluation of Orbital Volume
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Edward B. Strong, MD, University of California Davis
Other Study IDs: 200715801-1; IORG: 0000251
Record Dates: First submitted 2007-12-26; First posted 2008-01-02 (Estimated); Last update posted 2010-12-20 (Estimated); Status verified 2010-12

CONDITIONS: Orbital Fractures
Keywords: orbital fractures
MeSH Terms: conditions — Orbital Fractures

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
A retrospective review to assess the performance and clinical predictive value of a novel software program (Maxillo) designed to perform complex volumetric analysis with application in the field of orbital trauma.

DETAILED DESCRIPTION:
The concept of open reduction and internal fixation of large and complex traumatic orbital deformities is well established. It is known that successful orbital reconstruction hinges upon restoration of native orbital volume in order to establish pre-morbid function and avoid long-term complications. To date, a facile, reliable, and reproducible method to measure orbital volume has not been rendered, despite numerous approaches. The objective of this study is to assess the performance and clinical predictive value of a novel software program designed to perform complex volumetric analysis with application in the field of orbital trauma.

ELIGIBILITY:
Inclusion Criteria:

* Chart reviews of patients at UCDMC with orbital trauma and having operative repair of the orbital fractures with post-reduction imaging included.

Exclusion Criteria:

* Absences of post-operative imaging

Ages: 3 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with complex maxillofacial and orbital trauma that underwent operative repair of orbital fractures. Computer tomography scans from a cohort of patients with normal CT data sets will also be collected to assess "normative" orbital volumes.
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2007-11; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward B Strong, MD, Principal Investigator — University of California, Davis